CLINICAL TRIAL: NCT05232435
Title: Pilate Mat Exercise Versus Muscle Energy Technique on Chronic Non Specific Low Back Pain
Acronym: MET-LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hager Nazieh Mohamed Hekal, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002135
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Chronic Non Specific Low Back Pain
Keywords: LBP; Pilate mat exercise; MET

STUDY DESIGN:
Intervention Model Description: The trial has 3 groups
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pilate group (Experimental): will receive pilate exercise(1- bridging 2- shoulder bridge 3- front support 4- spine stretch forward 5- spine twist) and standard treatment (stretch hamstring , stretch lower back , strength abdominal muscles and electrical heat pad) for 12 sessions(3 sessions/week) over a period of four weeks.
  Interventions: Other: pilate mat exercise will be performed
- MET (Experimental): will receiveMET treatment for hamstring and erector spinae and standard treatment(stretch hamstring , stretch lower back , strength abdominal muscles and electrical heat pad) for 12 sessions (3 sessions/week)over a period of four weeks.
  Interventions: Other: MET
- control group (Active Comparator): will receive standard treatment(stretch hamstring , stretch lower back , strength abdominal muscles and electrical heat pad) only for 12 sessions (3 sessions/week) over a period of four weeks.
  Interventions: Other: control group receive standard treatment

INTERVENTIONS:
Other: pilate mat exercise will be performed — pilate group:1- bridging 2- shoulder bridge 3- front support 4- spine stretch forward 5- spine twist plus standard treatment(stretch hamstring -stretch lower back - strength abdominal muscles - electrical heat pad)
  Arms: pilate group
Other: MET — Will receive MET for hamstring and erectorspinae plus standard treatment
  Arms: MET
Other: control group receive standard treatment — electrical heat pad - stretch hamstring - stretch lower back muscles - stregth abdominal muscles
  Arms: control group

SUMMARY:
to investigate the effect of pilat mat exercise versus MET on chronic non specific LBP:Randomized controlled trial

DETAILED DESCRIPTION:
Low back pain (LBP) affects almost everyone at least once per life. Hence,it has been considered one of the most common musculoskeletal problems.The Pilates Method starts by strengthening the core, which is achieved by coordinating breathing with movement. Muscle energy technique is an associate degree of osteopathic manipulation methodology. The muscles of patients were used, on request, to type a singular controlled position, in a very specific direction, and against a distinctly executed therapist-applied counterforce.pilate mat exercise and muscle energy technique play a major role in treatment of patients with chronic non specific LBP so this trial will be conducted to investigate the effect of pilat mat exercise versus MET on chronic non specific LBP:

ELIGIBILITY:
Inclusion Criteria:

* Seventyeight Subjects will be selected from both genders, with age above 18 years.
* Normal body mass index (BMI) will be included.
* Participants diagnosed with chronic nonspecific LBP.

Exclusion Criteria:

* The participants will be excluded if they had one of the following criteria:
* Patient with previous back surgery, lumbar disc herniation, spinal deformities.
* Neuromusculoskeletal problems as hip arthrodesis or arthroplasty and spondylolisthesis.
* History of Cardiovascular disease, diabetes mellitus and rheumatoid arthritis
* Pregnant women and Osteoprosis.
* Leg length discrepancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-03-30 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to 4 weeks for each group
  using visual analogue scale.each patient willbe instructed to rate the current level of pain by placing (X) sign across the horizontal VAS line. The distance in millimeters from the lower limit was measured using a ruler. VAS will be assessed before and after the treatment program.as 1:2 mild , 3:6moderate and 7:10 sever pain.
functional disability | up to 4 weeks for each group
  using ronald morris questioneer.The RMDQ is scored by adding up the number of items the patient has ticked. Scores can vary between 0-24. Greater levels of disability are reflected by higher scores
ROM | up to 4 weeks for each group
  using BROMII.Use the two universal inclinometers to make flexion/extension measurements. Measurements with the universal inclinometer need to be with the patient in an upright position.
  1. Palpate and mark S1 and T12. Mark on bare skin when possible. This avoids the marks moving with the patient's clothing (Fig.2)
  2. Center the two inclinometers over the palpation marks and zero with your finger by spinning the dial (zero would then be at the bottom of the inclinometer).
  3. Have the patient flex forward as far as possible (Fig. 3). Note the reading on each inclinometer.
  4. The reading on the upper inclinometer is total lumbar flexion. The reading on the lower inclinometer is sacral flexion. The difference between the reading at S1 and T12 is true lumbar flexion.
  5. Repeat flexion protocol for extension having the patient extend back for full extension instead of flexing forward
flexibility | upto 4 weeks for each group
  using V sit and reach test.The test is done twice with a short break in between . Scoring: Zero point is at the level of feet. (We note negative values towards our body and positive values outward from our body.) The best trial is recorded in centimeters by best score

CONTACTS AND LOCATIONS:
Overall Officials: hager hekal, PHD student, Study Chair — faculty of physical therapy